CLINICAL TRIAL: NCT02063906
Title: Prognostic Relevance of Biological Subtype Overrides That of TNM Staging in Breast Cancer: Discordance Between Stage and Biology
Brief Title: Prognostic Relevance of Biological Subtype in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young-Hyuck Im, Professor, Samsung Medical Center
Other Study IDs: 2014-02-045
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer stage I-III: who received curative surgery for stage I-III breast cancer and had available data on immunohistochemistry profiles including hormone receptor status (HR) status, human epidermal growth factor receptor 2 (HER2) status, and Ki 67 staining at Samsung Medical Center from January 2004 to September 2008.

SUMMARY:
Recently, the investigators face "on the edges" for treatment decision to decide adjuvant systemic treatment, especially for patients who show discordance between stage and tumor biology. The aim of this study was to compare the prognostic relevance of the TNM staging system and intrinsic subtype in breast cancer patients who received curative surgery.

DETAILED DESCRIPTION:
Identified patients who received curative surgery for stage I-III breast cancer and had available data on immunohistochemistry profiles including hormone receptor status (HR) status, human epidermal growth factor receptor 2 (HER2) status, and Ki 67 staining at Samsung Medical Center from January 2004 to September 2008. Primary outcomes were recurrence-free survival (RFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* patients who received curative surgery
* stage I-III breast cancer
* between January 2004 and September 2008
* had available immunohistochemistry profiles.

exclusion Criteria:

* age <18 years old
* microinvasive carcinoma of breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received curative surgery for stage I-III breast cancer between January 2004 and September 2008 and had available immunohistochemistry profiles.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  was measured from the first date of diagnosis of breast cancer to the date of death or the last follow-up visit

SECONDARY OUTCOMES:
Recurrence-free survival | 1 Year
  was defined as the time from the date of curative resection to the date when breast cancer recurred, irrespective of locoregional recurrences including ipsilateral and contralateral breast recurrences or distant metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hyuck Im, Pf, Principal Investigator — Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea